CLINICAL TRIAL: NCT05248308
Title: Genicular Artery Embolization (GAE) for the Treatment of Chronic Post Knee Arthroplasty Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Fundings challenges
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Yan Epelboym, M.D.,M.P.H., Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000238
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Knee Pain Chronic; Knee Swelling Pain; Arterial Occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Genicular artery embolization (Experimental): Study participants will undergo genicular artery embolization (GAE) for treatment of chronic moderate to severe pain following knee arthroplasty or revision arthroplasty. Embolization will be performed using Embozene Microspheres.
  Interventions: Device: Embozene Microspheres

INTERVENTIONS:
Device: Embozene Microspheres — Embozene Microspheres are manufactured by Varian Medical Systems (Palo Alto, CA). These microspheres are non-resorbable hydrogel microspheres coated with polyzene-F. Embozene microspheres are approved for use in treating arteriovenous malformations, hypervascular tumors such as uterine fibroids and hepatomas, and prostatic arteries in patients with benign prostatic hyperplasia.
  One of the causes of chronic pain in the setting of a knee arthroplasty may be increased blood flow to the specific area(s) of pain. The purpose of this procedure is to reduce blood flow (embolize) to specific parts of the knee which are contributing to your pain.
  This procedure is performed by infusing the Embozene particles into specific knee arteries (genicular arteries) in the region of knee pain.

SUMMARY:
This study seeks to evaluate the safety and efficacy of genicular artery embolization (GAE) as a treatment for patients with chronic pain following primary total knee arthroplasty (TKA) or revision TKA at 6 months as measured by the Knee Injury and Osteoarthritis Outcome Score (KOOS).

DETAILED DESCRIPTION:
This is a single center, single arm, prospective pilot study evaluating the safety and efficacy of genicular artery embolization (GAE) for treatment of chronic pain following primary total knee arthroplasty (TKA) or revision TKA. Following screening, eligible participants will be offered enrollment. Patients who demonstrate baseline imaging findings of knee synovitis either on US, MRI, or both modalities will be offered GAE. Genicular artery embolization will be performed using a SeQure® microcatheter (Guerbet LLC, Villepinte, France) using Embozene microspheres (Varian Medical Systems, Palo Alto, CA).

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory
2. History of total knee arthroplasty or revision arthroplasty in the symptomatic knee
3. Moderate to severe knee pain: pain VAS ≥50 mm
4. Knee pain resistant to at least 3 months of conservative therapy including pharmacologic therapy or intra-articular injection.
5. Absence of pregnancy at time of screening as determined by urine HCG
6. Provision of signed and dated informed consent form
7. Willing, able, and mentally competent to provide informed consent and to tolerate angiography, US, and MRI.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of severe peripheral arterial disease symptoms including claudication, diminished or absent lower extremity pulses, leg numbness or weakness or known arterial atherosclerosis or occlusion that would limit selective angiography
2. History of inflammatory arthropathy such as rheumatoid arthritis, spondyloarthropathies, crystal disease, gout, pseudogout, or lupus
3. Presence of non-MRI compatible devices (e.g., cardiac pacemaker).
4. Known history of anaphylaxis to iodinated or gadolinium-based contrast agents
5. BMI greater than 50
6. Renal dysfunction as defined by serum creatinine >1.6 dl/mg or eGFR <60 obtained within 30 days of procedure.
7. Uncorrectable coagulopathy (platelet count < 50,000, international normalized ratio >1.5 within 30 days of procedure
8. Active systemic or local knee infection
9. Pregnant or intent to become pregnant during the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
KOOS - Pain subscale KOOS Scale - Pain | 6 months
  Estimate the effect of genicular artery embolization on the change in knee pain, as assessed by the KOOS, at 6 months post vs. pre-intervention, in patients with chronic knee pain following TKA

SECONDARY OUTCOMES:
VAS Scale | 6 months
  Estimate the effect of genicular artery embolization on the change in knee pain, as assessed by the VAS scale, at 1 week, 1, 3, and 6 months, in patients in patients with chronic knee pain following TKA.
Analgesic Utilization | 6 months
  Estimate the effect of genicular artery embolization on analgesic utilization as measured by morphine equivalents and non-steroidal anti-inflammatories utilization
KOOS - Non-Pain Components | 6 months
  Estimate effect in non-pain components of the KOOS score (KOOS Symptoms, KOOS ADL, KOOS Sport ADL, and KOOS QOL) by comparing these scores at 1 week, 1,3, and 6 months to the pre-procedure score.
MHI-5 | 6 months
  Assess for associations between mental health and post TKA pain as assessed by the MHI-5 by comparing scores at 1 week, 1, 3, and 6 months to the pre-procedure score.
CRP & IL-6 | 6 months
  Estimate the effect of genicular artery embolization on CRP and IL-6, by comparing baseline laboratory values to 6-month post procedure values.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Epelboym, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States